CLINICAL TRIAL: NCT04627337
Title: Efficacy and Safety of Saccharomyces Boulardii CNCM I-745 in the Treatment of Small Intestinal Bacterial Overgrowth in Patients Suffering From Irritable Bowel Syndrome With Diarrhea
Brief Title: Efficacy and Safety of Saccharomyces Boulardii in the Treatment of Small Intestinal Bacterial Overgrowth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Principal Investigator, Juan Lasa, Clinical Professor, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIBO01
Record Dates: First submitted 2018-11-28; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saccharomyces boulardii (1 capsule of 250 ug BID) + Dietary advice (Experimental): Patients received 1 capsule of Saccharomyces boulardii 250 ug BID plus dietary advice for 15 days. Dietary advice consisted of a low fermentation diet which was delivered as a written list of food and beverages that patients should avoid adapted to local habits and an oral explanation by a health professional.
  Interventions: Drug: Saccharomyces Boulardii 250 MG; Behavioral: Dietary advice following a low fermentation diet
- Dietary advice without medication (Active Comparator): Patients received dietary advice for 15 days. Dietary advice consisted of a low fermentation diet which was delivered as a written list of food and beverages that patients should avoid adapted to local habits and an oral explanation by a health professional.
  Interventions: Behavioral: Dietary advice following a low fermentation diet

INTERVENTIONS:
Drug: Saccharomyces Boulardii 250 MG — Probiotic yeast in capsules
  Other Names: Dietary advice following a low fermentation diet
  Arms: Saccharomyces boulardii (1 capsule of 250 ug BID) + Dietary advice
Behavioral: Dietary advice following a low fermentation diet — Medical advice was delivered to patients to follow a low fermentation diet. A list of food and beverages to avoid was delivered along with specified instructions provided by a health professional

SUMMARY:
Non-constipated irritable bowel syndrome is a common disorder that may be related to small intestinal bacterial overgrowth. Saccharomyces boulardii CNCM I-745 is a probiotic yeast that has proven efficacy for the treatment of acute gastroenteritis and antibiotic-associated diarrhea. However, its efficacy for the treatment of diarrhea-predominant irritable bowel syndrome with small intestinal bacterial overgrowth has not been assessed. Hence, an exploratory randomized, open label trial comparing the efficacy and safety of Saccharomyes boulardii CNCM I-745 plus diet administration versus diet administration only for 15 days among adult patients with the aforementioned condition was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Diagnosis of Irritable Bowel syndrome according to Rome III criteria
* Diagnosis of concomitant small intestinal bacterial overgorwth (SIBO) by breath test

Exclusion Criteria:

* Pregnancy
* Diagnosis of Celiac disease
* Diagnosis of Inflammatory Bowel Disease or other immune-mediated gastrointestinal conditions
* Immunosuppression
* Diagnosis of active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity measured by the Irritable Bowel Syndrome Symptom Severity Scale | 15 days
  The IBS Symptom Severity Scale (IBS-SSS) is a validated questionnaire (Francis et al. 1997) that evaluates the intensity of the following IBS symptoms: abdominal pain, distension, stool frequency and consistency, and general impact on life. The IBS-SSS calculates the sum of these 5 items (each scored on a visual analogue scale from 0 to 100) and the score values range from 0 to 500 (maximum severity). An IBS-SSS questionnaire was filled-in by each randomized patient at both visits. We compared the difference between the overall score before and after the intervention.

SECONDARY OUTCOMES:
Change in hydrogen excretion measured by lactulose breath test | 15 days
  Presence of bacterial overgrowth was examined by a lactulose hydrogen breath test (LHBT), which measures hydrogen concentration within the expelled breath.
  Patients ingested 10 mL lactulose, then breath samples were collected every 20 minutes over 180 min and analyzed to determine hydrogen concentration. An excreted hydrogen concentration/time area under the curve (AUC) was then calculated. A positive test corresponded to any of the following results: rise in breath hydrogen at least 20 ppm above basal levels within 100 minutes after ingestion of lactulose; rise at least 12 ppm within100 minutes with a decrease of 5 ppm (markers of SIBO) and subsequent increase; (AUC) value of more than 3000 ppm. Changes in terms of absolute hydrogen excretion measured by AUC of hydrogen excretion over time were compared before and after intervention in every patient.

CONTACTS AND LOCATIONS:
Locations (1):
- CEMIC, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No